CLINICAL TRIAL: NCT05111730
Title: Effect of Shock Wave In Reducing Chemotherapy- Induced Peripheral Neuropathy In Adult and Pediatric Tumors Patients:A Randomized Controlled Trail
Brief Title: Effect of Shock Wave In Reducing Chemotherapy- Induced Peripheral Neuropathy In Adult and Pediatric Tumors Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed E. Ali, Ph. D Candidate., Assistant Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002568
Record Dates: First submitted 2021-10-13; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Peripheral Neuropathy
Keywords: PERIPHERAL NEUROPATHY; CHEMOTHERAPY; SHOCKWAVE
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Eighty children with tumors were enrolled in this study and were assessed for eligibility. Their aged ranged from eight and forty years. They were assigned randomly into two equal groups. Group (A) study group received the same medical care and shock wave, three times / weak for three successful months. And group (B) control group received medical care and standard chemotherapy only.Nerve conduction studies (NCS) and somatosensory-evoked potentials (SSEPs) were used to assess peripheral neuropathy pre and post intervention. All children were assisted before and after three months of intervention.
Who Masked: Outcomes Assessor
Masking Description: Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group A (study group) and Group B ( control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The shockwave Group (Experimental): Group (A) study group received medical care and standard chemotherapy and shock wave, three times / week for three successful months.
  Interventions: Device: The Shock wave Therapy.
- the traditional treatment group (No Intervention): group (B) control group received medical care and standard chemotherapy only.

INTERVENTIONS:
Device: The Shock wave Therapy. — Shockwave therapy is a multidisciplinary device used in orthopedics, physiotherapy, sports medicine, urology and veterinary medicine. Its main assets are fast pain relief and mobility restoration. Together with being a non-surgical therapy with no need for painkillers makes it an ideal therapy to speed up recovery and cure various indications causing acute or chronic pain. Shockwave is an acoustic wave which carries high energy to painful spots and myoskeletal tissues with sub-acute, sub-chronic and chronic conditions. The energy promotes regeneration and reparative processes of the bones, tendons and other soft tissues. Shockwaves are characterized by jump change in pressure, high amplitude and non-periodicity. The kinetic energy of the projectile, created by compressed air, is transferred to the transmitter at the end of the applicator and further into the tissue.
  Arms: The shockwave Group

SUMMARY:
This study aimed to assess the efficacy of shock wave in reducing Chemotherapy- Induced Peripheral Neuropathy in adult and pediatric tumors patients.

DETAILED DESCRIPTION:
Peripheral neuropathy is a serious condition characterized by symmetrical, distal damage to the peripheral nerves that may be caused by several classes of drugs, including chemotherapeutic agents. Chemotherapy-induced peripheral neuropathy (CIPN) is an adverse effect estimated to occur in up to 40% of patients undergoing chemotherapy, with its incidence increasing in patients being treated with multiple agents. Pharmacists play a pivotal role in the prevention and management of CIPN by recommending evidence-based pharmacologic and nonpharmacologic strategies appropriate for the individual patient.Peripheral neuropathy (PN) is a systemic disease characterized by symmetrical, distal damage to the peripheral nerves that negatively impacts patient quality of life (QOL). Prolonged symptoms associated with PN can cause pain, interfere with functional ability (e.g., dressing, driving, house-work), and disrupt emotional health.

ELIGIBILITY:
Inclusion Criteria:

* Their age will ranging from eight to forty years.
* All cases participated in this study will from both sexes.
* All cases receiving chemotherapy as primary treatment, postoperative surgical removal of tumors or with conjunction with radiotherapy
* All cases have polyneuropathy caused by chemotherapy.

Exclusion Criteria:

* Patient with osteoporosis.
* Patient with DVT.
* Patient have a Pacemaker fitted
* Uncooperative patients

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Malondialdehyde (MDA) as oxidative stress marker | Malondialdehyde (MDA) level was assessed at day 0.
  Malondialdehyde level in blood will be measured
Malondialdehyde (MDA) as oxidative stress marker | Malondialdehyde (MDA) level will be assessed at day 90.
  Malondialdehyde level in blood will be measured
Interlukin 6 (IL-6) as inflammatory marker | Interlukin 6 (IL-6) level was assessed at day 0.
  Interlukin 6 (IL-6) level in blood will be measured
Interlukin 6 (IL-6) as inflammatory marker | Interlukin 6 (IL-6) level will be assessed at day 90.
  Interlukin 6 (IL-6) level in blood will be measured
Plasma Neurotensin (NT) as potential marker for neuropathic pain | Plasma Neurotensin (NT)level was assessed at day 0.
  Plasma Neurotensin (NT) level in blood will be measured
Plasma Neurotensin (NT) as potential marker for neuropathic pain | Plasma Neurotensin (NT)level will be assessed at day 90.
  Plasma Neurotensin (NT) level in blood will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed E Ali, Ph.D student, Principal Investigator — South Valley University
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No